CLINICAL TRIAL: NCT06898671
Title: Language Outcomes, Mechanisms, and Trajectories in Adults With and Without Developmental Language Disorder
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Kristi I. Hendrickson, Assistant Professor, University of Iowa
Other Study IDs: 202204590; 1R01DC020143-01 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Developmental Language Disorder
Keywords: Language Profiles; Language Processing; Adult Language Disorders; Typical Adult Language
MeSH Terms: conditions — Language Development Disorders; Language Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Developmental Language Disorder: Adults with below average language skills participate in eye tracking tasks
  Interventions: Behavioral: Eye-Tracking in Visual World Paradigm
- Typically Developing: Adults with typical language skills participate in eye tracking tasks
  Interventions: Behavioral: Eye-Tracking in Visual World Paradigm

INTERVENTIONS:
Behavioral: Eye-Tracking in Visual World Paradigm — Participants complete six eye tracking tasks. They see images on a computer screen are tasked with finding a specific picture or saying a specific word (target). We track their eye movements to the visual representations of the target compared with their eye movements to visual representations of items that are similar to the target.

SUMMARY:
The investigators' overall objective is to characterize the long-term outcomes of Developmental Language Disorder (DLD) in adulthood and to identify specific cognitive mechanisms mediating these outcomes. To address their objectives, the investigators utilize a large, pre-existing dataset and participant pool from one of the most comprehensive examinations of DLD to date: the Iowa Longitudinal Study. The investigators will re-recruit subjects with DLD and with typical language from this historic cohort, who are now adults (30-35 years old). In Aim 1, the investigators will use measures from kindergarten through 10th grade and collect new outcome measures in adulthood to characterize the long-term outcomes of DLD. The investigators predict that adults with DLD will diverge from adults with TL in language skills that are more complex and higher-level language skills that are important for communication in the workplace. Further, the investigators predict a fanning effect: some children with DLD will "catch up" to their TL peers in adulthood, some will show evidence of a decline, and others will show stable trajectories. In Aim 2, the investigators measure real-time competition across written and spoken language using eye-tracking. According to speed of processing accounts adults with DLD may be slower than their TL peers to activate competitors and targets. According to working memory accounts adults with DLD will show sustained competitor activation. Further, the investigators predict that measures related to the dynamics of competition (speed of activation and timing of competitor suppression) will account for variation in language outcomes in adults.

DETAILED DESCRIPTION:
Aim 1: Characterize individual differences in the developmental trajectory and ultimate attainment of language ability in adults with and without DLD. This proposal directly addresses previous limitations by leveraging existing data and an existing participant pool from one of the most unique, influential, and comprehensive examinations of childhood DLD to date (the Iowa Longitudinal Study). The investigators re-recruit participants with and without DLD from this historic study who are now adults (30-35 years old). The investigators use retrospective oral language measures from kindergarten through 10th grade and collect new measures that capture language comprehensively (receptive and expressive language at the sublexical, lexical, sentence, and discourse/pragmatic levels) in adulthood. The investigators focus on the following two sub-aims:

Aim 1a: Characterize language outcomes in adults with DLD. The proposed measures will capture language abilities that stratify a wide range of language skills in adolescents and adults, differentiate individuals with DLD from their typically developing peers at various stages of development, and are reported to be functional for adults in the workplace. Given documented difficulties with complex language structures and discourse in older children and adolescents with DLD, the investigators expect that adults with DLD may diverge from adults with TL in performance related to language skills that are more linguistically complex (e.g., complex syntax and high lexical density). Further, they predict marked deficits in higher-level language skills (pragmatics and discourse), which are important aspects of communication in the workplace (e.g., language used for negotiating, cooperating, etc.). Given variable profiles of DLD, the investigators also expect that some participants will demonstrate lingering differences related to the consistency of their errors and the phonological complexity of their utterances. The investigators also seek to answer questions about the dimensionality of language ability. This follows from previous work demonstrating that language ability is best captured by a unitary factor in the early school-age years, with vocabulary and grammar becoming differentiated only later in development. Accordingly, the investigators carry out analyses to determine whether this dual-factor approach holds in adulthood or whether the dimensionality has increased yet further, and whether differences in language dimensionality obtain across DLD and TL groups.

Aim 1b: Shape of developmental trajectory. The investigators use retrospective language measures collected from K-10th grade as part of the Iowa Longitudinal Study, combined with new measures the investigators will collect in these same individuals in adulthood to examine the long-term trajectory of DLD. Given that adults with DLD do not typically receive services, the status quo under which the field is implicitly operating is that adults with DLD "catch-up" to their TL peers or that language abilities plateau in the school-age years and no further development is possible. However, research shows that adults with DLD have lower quality of life outcomes, and language abilities continue to grow until the thirties in typical populations, which conflicts with this viewpoint. For this sub-aim, the investigators use latent-trait Bayesian analyses to mediate between two competing hypotheses. The first hypothesis is that the investigators will uncover evidence for the maintenance of the relative stability seen during the school-age years (i.e., children, with remarkable reliability, maintain their standing relative to the rest of the cohort members in longitudinal studies of language ability). However, upon exiting the educational system, adults with DLD rarely receive services, and this may contribute to increased variability in outcomes. Thus, the second, competing hypothesis is that the investigators will uncover a fanning effect: some adults will have improved their language abilities relative to their prior standing in the cohort, while others will show evidence of a decline, with still others showing a relative maintenance of the school-age years trajectory. Such a fanning effect would suggest that trajectories after the school-age years are amenable to intervention.

Aim 2: Identify real-time processes that explain individual differences in language outcomes in adults with and without DLD.

For Aim 2, the investigators offer a mechanistic account of language deficits underlying DLD in adults. Their goal is to refine processing-based theories of DLD by offering a more precise characterization of the computational differences that subserve deficits in language processing in this population. Further, the investigators seek to illuminate individual differences in adult language across the ability spectrum. For this aim, the investigators use well supported models of competition in adults with TL as a theoretical framework for understanding mechanisms that underlie language deficits in adults with DLD. The investigators have developed a research protocol that measures real-time competition in expressive and receptive language at the lexical, sentence, and pragmatic levels. Consistent with working memory accounts, the investigators predict that, compared to adults with TL, adults with DLD will show sustained competition at all levels of language. An alternative-though not mutually exclusive- hypothesis is consistent with speed of processing accounts: group differences will be better reflected in how quickly targets and competitors are initially activated. Further, the investigators predict that measures related to the dynamics of competition will account for variation in language outcomes in adults across the ability spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Developmental Language Disorder (DLD) and those with typical language (TL) between the ages of 28 and 40 years who participated in the Iowa Longitudinal Study(NIH-DC-19-90 & P50 DC002746; IRB# 200106051, "Collaboration on Specific Language Impairment".)
* Aged 30-35
* Normal or corrected to normal vision
* Normal hearing

Exclusion Criteria:

* history of brain injury
* history of neural developmental disabilities
* not monolingual

Ages: 30 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 150 adults with Developmental Language Disorder (DLD) and 250 adults with typical language (TL) will participate in this project. Participants will be between the ages of 30 and 34 years at time of enrollment. Participants will be drawn from a large cohort of adults with and without DLD who participated in the Iowa Longitudinal Study (an extensive longitudinal follow-up of an epidemiological study of DLD)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Eye movements | 2 hours
  Participant are presented with images, and here words referring two one of the images while their eye movements are tracked. We measure the proportion fixations to the target image and distractor images over time. The measurement tool we are using is an eye-tracker (EyeLink portable duo)
  Note this is BESH, no intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stewart McCauley, PhD, Principal Investigator — University of Iowa; Si On Yoon, PhD, Principal Investigator — University of Iowa; Philip Combiths, PhD, Principal Investigator — University of Iowa; J. Bruce Tomblin, PhD, Principal Investigator — University of Iowa; Jacob Oleson, PhD, Principal Investigator — University of Iowa
Locations (1):
- Wendell Johnson Speech and Hearing Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected from this project will be used only for research and educational purposes.
  Our proposed research will achieve scientific rigor as defined by NIH. Both experimental details and data will be available to achieve transparency:
  1. We will make the detailed procedure of experiments available to other researchers so that the results can be reproduced across different laboratories
  2. We will also have the deidentified data (both subject and item level) that protects subject confidentiality posted to the PI's lab website or Co-I's lab Open Science Framework (OSF) website as the results are published, and
  3. All statistical models used in the published papers will be posted to the PI's lab website or Co-I's lab OSF website.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared upon the conclusion of the project without an end date
Access Criteria: 1. We will make the detailed procedure of experiments available to other researchers so that the results can be reproduced across different laboratories
  2. We will also have the deidentified data (both subject and item level) that protects subject confidentiality posted to the PI's lab website or Co-I's lab Open Science Framework (OSF) website as the results are published, and
  3. All statistical models used in the published papers will be posted to the PI's lab website or Co-I's lab OSF website.

DOCUMENTS (1):
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT06898671/ICF_000.pdf